CLINICAL TRIAL: NCT05606874
Title: Retention Rate and Caries Preventive Effect of Preheated Flowable Resin Composite Used as a Pit and Fissure Sealant Versus Conventional Resin-based Fissure Sealant in Patients With Permanent Molars With Deep Pit and Fissure Over One Year Follow up. A Randomized Clinical Trial
Brief Title: Retention Rate and Caries Preventive Effect of Preheated Flowable Resin Composite Used as a Pit and Fissure Sealant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, safa abd alwahab natiq, operator, data entry and corresponding author; B.D.S. Cairo University (2016), Conservative Dentistry Department, Faculty of Dentistry, Cairo University. Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: preheated flowable composite
Record Dates: First submitted 2022-10-29; First posted 2022-11-07 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2022-03

CONDITIONS: Pit and Fissure Sealant
Keywords: preheated flowable composite; pit and fissure sealant; Retention Rate
MeSH Terms: conditions — Van der Woude syndrome | interventions — Pit and Fissure Sealants; Ultra Seal XT

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-heating of flowable resin composite . (Experimental): (Filtek™ Z350Xt Flowable Restorative, 3M ESPSE, USA)
  Interventions: Other: Pre-heating of flowable resin composite used as a pit and fissure sealant.
- Conventional resin fissure sealant (Active Comparator): (total etch), (UltraSeal XT®, Ultradent, USA)
  Interventions: Other: Conventional resin fissure sealant

INTERVENTIONS:
Other: Pre-heating of flowable resin composite used as a pit and fissure sealant. — The occlusal fissures will be etched with a 37% phosphoric acid gel for 30 s. After rinsing the enamel with water for 30 s the enamel will be dried for 15 s with compressed air. After completing the fissure preparations a single coat of adhesive (3M ESPE ADPER ,USA) will be applied to the etched surface ,dried under gentle air flow for 2- 3 s and light cured for 20 s using a LED light curing unit with a 1000 mw output .Conventional resin fissure sealant (total etch), (UltraSeal XT®, Ultradent, USA) will be applied to the etched pits and fissures. After removing the rubber dam the occlusion will be checked the sealant will be adjusted with a composite finishing bur and polished with polishing points.
  Other Names: (Filtek™ Z350Xt Flowable Restorative, 3M ESPSE, USA)
  Arms: Pre-heating of flowable resin composite .
Other: Conventional resin fissure sealant — The occlusal fissures will be etched with a 37% phosphoric acid gel for 30 s. After rinsing the enamel with water for 30 s the enamel will be dried for 15 s with compressed air. After completing the fissure preparations a single coat of adhesive (3M ESPE ADPER ,USA) will be applied to the etched surface ,dried under gentle air flow for 2- 3 s and light cured for 20 s using a LED light curing unit with a 1000 mw output .Conventional resin fissure sealant (total etch), (UltraSeal XT®, Ultradent, USA) will be applied to the etched pits and fissures. After removing the rubber dam the occlusion will be checked the sealant will be adjusted with a composite finishing bur and polished with polishing points.
  Other Names: (total etch), (UltraSeal XT®, Ultradent, USA)
  Arms: Conventional resin fissure sealant

SUMMARY:
Retention rate and caries preventive effect of preheated flowable resin composite used as a pit and fissure sealant versus conventional resin-based fissure sealant in patients with permanent molars with deep pit and fissure over one year follow up. A randomized clinical trial

DETAILED DESCRIPTION:
Statement of the problem:

Pit and fissure sealant placement is considered as an effective modality for prevention of caries on occlusal surfaces. Penetration, retention and lateral wall adaptation are the key factors in success of pit and fissure sealant restorations .

The retention is very critical for the sealing material and the successful penetration of the material into the pits and fissures However, the morphology of the fissures significantly influences the penetration of the sealing material occlusal fissure pattern like in deep and narrow fissures like I-type and IK- type where lesser penetration may be encountered fillers are added to the pit and fissure sealants in order to increase their wear and abrasion resistance. However, these fillers could lead to increase in the viscosity with subsequent decrease in the penetration.

Rationale:

According to a systematic review, they found that preheating of resin composite apparently increases the flowability of regular consistency composites, which improves the adaptation of the material into the cavity walls. Also studied the effect of heat and sonic vibration on penetration of flowable resin composite, they found that higher penetration was associated with heat compared with the conventional application method. So, this proposal is introduced with the hypothesis that preheating of filled fissure sealants may enhance their flowability and penetration especially into those fissures with complex structure.

ELIGIBILITY:
Inclusion Criteria:

participant:

1. Young adults (16_22y)
2. Patients who have existing pits and fissures that are anatomically deep and caries susceptible.

Teeth

1. Permanent molars teeth without any caries and cavitation. (Azarpazhooh & Main 2008)
2. Permanent molar teeth that have deep pit and fissure morphology, with "sticky" fissures.
3. Permanent molar teeth with stained grooves.
4. Stained pits and fissures with minimum decalcification of opacification and no softness at the base of the fissure (ICDAS 1 and 2).

   -

Exclusion Criteria:

participant:

1. Uncooperative behavior, limits the use of sealants due to hampering of adequate field or isolation techniques throughout the procedure.
2. Patients allergic to sealant material.
3. Patient with history of medical disease, drug therapies or any other serious relevant problem.

Teeth:

1. An individual with no previous caries experience and well coalesced pits and fissures
2. Partially erupted teeth.
3. Teeth with cavitation or caries of the dentin.
4. A large restoration is present on occlusal surface.
5. If pits and fissures are self-cleansable.
6. Teeth with dental fluorosis, hypocalcification or hypercalcification

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Retention rate | T1: 3 months
  Retention criteria
Retention rate | T2: 6 months
  Retention criteria
Retention rate | T3: 12 months
  Retention criteria

SECONDARY OUTCOMES:
Caries incidence | T1: 3 months
  ICDAS-II visual criteria
Caries incidence | T2: 6 months
  ICDAS-II visual criteria
Caries incidence | T3: 12 months
  ICDAS-II visual criteria

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abouauf, Ass.prof, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Featherstone JD. Dental caries: a dynamic disease process. Aust Dent J. 2008 Sep;53(3):286-91. doi: 10.1111/j.1834-7819.2008.00064.x. PMID 18782377
- [Background] Erbas Unverdi G, Atac SA, Cehreli ZC. Effectiveness of pit and fissure sealants bonded with different adhesive systems: a prospective randomized controlled trial. Clin Oral Investig. 2017 Sep;21(7):2235-2243. doi: 10.1007/s00784-016-2016-8. Epub 2016 Nov 30. PMID 27900529
- [Background] Subramaniam P, Konde S, Mandanna DK. Retention of a resin-based sealant and a glass ionomer used as a fissure sealant: a comparative clinical study. J Indian Soc Pedod Prev Dent. 2008 Sep;26(3):114-20. doi: 10.4103/0970-4388.43192. PMID 18923223
- [Background] Rickman LJ, Padipatvuthikul P, Chee B. Clinical applications of preheated hybrid resin composite. Br Dent J. 2011 Jul 22;211(2):63-7. doi: 10.1038/sj.bdj.2011.571. PMID 21779058
- [Background] Ramesh H, Ashok R, Rajan M, Balaji L, Ganesh A. Retention of pit and fissure sealants versus flowable composites in permanent teeth: A systematic review. Heliyon. 2020 Sep 24;6(9):e04964. doi: 10.1016/j.heliyon.2020.e04964. eCollection 2020 Sep. PMID 33005790
- [Background] Nahvi A, Razavian A, Abedi H, Charati JY. A comparison of microleakage in self-etch fissure sealants and conventional fissure sealants with total-etch or self-etch adhesive systems. Eur J Dent. 2018 Apr-Jun;12(2):242-246. doi: 10.4103/ejd.ejd_63_18. PMID 29988227
- [Background] Lopes LCP, Terada RSS, Tsuzuki FM, Giannini M, Hirata R. Heating and preheating of dental restorative materials-a systematic review. Clin Oral Investig. 2020 Dec;24(12):4225-4235. doi: 10.1007/s00784-020-03637-2. Epub 2020 Oct 20. PMID 33083851
- [Background] Khare M, Suprabha BS, Shenoy R, Rao A. Evaluation of pit-and-fissure sealants placed with four different bonding protocols: a randomized clinical trial. Int J Paediatr Dent. 2017 Nov;27(6):444-453. doi: 10.1111/ipd.12281. Epub 2016 Dec 26. PMID 28024165
- [Background] Kim HJ, Choi HJ, Kim KY, Kim KM. Effect of Heat and Sonic Vibration on Penetration of a Flowable Resin Composite Used as a Pit and Fissure Sealant. J Clin Pediatr Dent. 2020;44(1):41-46. doi: 10.17796/1053-4625-44.1.7. PMID 31995416
- [Background] Jafarzadeh M, Malekafzali B, Tadayon N, Fallahi S. Retention of a Flowable Composite Resin in Comparison to a Conventional Resin-Based Sealant: One-year Follow-up. J Dent (Tehran). 2010 Winter;7(1):1-5. Epub 2010 Mar 31. PMID 21998768
- [Background] Irinoda Y, Matsumura Y, Kito H, Nakano T, Toyama T, Nakagaki H, Tsuchiya T. Effect of sealant viscosity on the penetration of resin into etched human enamel. Oper Dent. 2000 Jul-Aug;25(4):274-82. PMID 11203831
- [Background] Ganesh M, Shobha T. Comparative evaluation of the marginal sealing ability of Fuji VII and Concise as pit and fissure sealants. J Contemp Dent Pract. 2007 May 1;8(4):10-8. PMID 17486182
- [Background] Rishika, Garg N, Mayall SS, Pathivada L, Yeluri R. Combined Effect of Enamel Deproteinization and Intermediate Bonding in the Retention of Pit and Fissure Sealants in Children: A Randomized Clinical Trial. J Clin Pediatr Dent. 2018;42(6):427-433. doi: 10.17796/1053-4625-42.6.4. Epub 2018 Aug 7. PMID 30085876
- [Background] Garg N, Indushekar KR, Saraf BG, Sheoran N, Sardana D. Comparative Evaluation of Penetration Ability of Three Pit and Fissure Sealants and Their Relationship with Fissure Patterns. J Dent (Shiraz). 2018 Jun;19(2):92-99. PMID 29854882
- [Background] Erdemir U, Sancakli HS, Yaman BC, Ozel S, Yucel T, Yildiz E. Clinical comparison of a flowable composite and fissure sealant: a 24-month split-mouth, randomized, and controlled study. J Dent. 2014 Feb;42(2):149-57. doi: 10.1016/j.jdent.2013.11.015. Epub 2013 Dec 1. PMID 24296163
- [Background] Dukic W, Dukic OL, Milardovic S, Vindakijevic Z. Clinical comparison of flowable composite to other fissure sealing materials--a 12 months study. Coll Antropol. 2007 Dec;31(4):1019-24. PMID 18217452
- [Background] Bagherian A, Shirazi AS. Flowable composite as fissure sealing material? A systematic review and meta-analysis. Br Dent J. 2018 Jan 26;224(2):92-97. doi: 10.1038/sj.bdj.2018.40. PMID 29372708
- [Background] Aman N, Khan FR, Salim A, Farid H. A randomized control clinical trial of fissure sealant retention: Self etch adhesive versus total etch adhesive. J Conserv Dent. 2015 Jan-Feb;18(1):20-4. doi: 10.4103/0972-0707.148883. PMID 25657521
- [Background] Oba AA, Sonmez IS, Ercan E, Dulgergil T. Comparison of retention rates of fissure sealants using two flowable restorative materials and a conventional resin sealant: two-year follow-up. Med Princ Pract. 2012;21(3):234-7. doi: 10.1159/000333561. Epub 2011 Dec 8. PMID 22156663
- [Background] Beun S, Bailly C, Devaux J, Leloup G. Physical, mechanical and rheological characterization of resin-based pit and fissure sealants compared to flowable resin composites. Dent Mater. 2012 Apr;28(4):349-59. doi: 10.1016/j.dental.2011.11.001. Epub 2011 Nov 25. PMID 22119547
- [Background] Aguilar FG, Drubi-Filho B, Casemiro LA, Watanabe MG, Pires-de-Souza FC. Retention and penetration of a conventional resin-based sealant and a photochromatic flowable composite resin placed on occlusal pits and fissures. J Indian Soc Pedod Prev Dent. 2007 Oct-Dec;25(4):169-73. doi: 10.4103/0970-4388.37012. PMID 18007102